CLINICAL TRIAL: NCT01395810
Title: Safety and Efficacy of NNC-0156-0000-0009 After Long-Term Exposure in Patients With Haemophilia B
Brief Title: Safety and Efficacy of NNC-0156-0000-0009 After Long-Term Exposure in Patients With Haemophilia B: An Extension to Trials NN7999-3747 and NN7999-3773
Acronym: paradigm™ 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN7999-3775; 2010-023072-17 (EudraCT Number); U1111-1121-5408 (Other: WHO); JapicCTI-121812 (Registry Identifier: JAPIC)
Record Dates: First submitted 2011-06-30; First posted 2011-07-18 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: Congenital Bleeding Disorder; Haemophilia B
MeSH Terms: conditions — Hemophilia B | interventions — nonacog beta pegol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Prophylaxis, high dose (once weekly) (Experimental)
  Interventions: Drug: nonacog beta pegol
- Prophylaxis, low dose (once weekly) (Experimental)
  Interventions: Drug: nonacog beta pegol
- On-demand (Experimental)
  Interventions: Drug: nonacog beta pegol
- Prophylaxis, high dose (every second week) (Experimental)
  Interventions: Drug: nonacog beta pegol

INTERVENTIONS:
Drug: nonacog beta pegol — One single dose administered intravenously (into the vein) once weekly. Patients will receive instruction on how to treat any bleeding episode they may experience.
  Other Names: NNC-0156-0000-0009
  Arms: Prophylaxis, high dose (once weekly); Prophylaxis, low dose (once weekly)
Drug: nonacog beta pegol — One single dose administered intravenously (into the vein). Patients will treat themselves with either a low or a high dose dependent on the severity of the bleeding episode.
  Other Names: NNC-0156-0000-0009
  Arms: On-demand
Drug: nonacog beta pegol — One single dose administered intravenously (into the vein) every second week. Patients will receive instruction on how to treat any bleeding episode they may experience.
  Other Names: NNC-0156-0000-0009
  Arms: Prophylaxis, high dose (every second week)

SUMMARY:
This trial is conducted in Asia, Europe, Japan, North America and South Africa. The aim is to evaluate the safety and efficacy of nonacog beta pegol (NNC-0156-0000-0009) after long-term exposure in patients with haemophilia B.

This trial is an extension to trials NN7999-3747 (NCT01333111/paradigm™ 2) and NN7999-3773 (NCT01386528/paradigm™ 3).

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in NN7999-3747 (NCT01333111) and/or NN7999-3773

Exclusion Criteria:

* Known history of FIX inhibitors based on existing medical records, laboratory report reviews and patient and LAR (legal acceptable representative) interviews
* Current FIX inhibitors above or equal to 0.6 BU (Bethesda Units)
* Congenital or acquired coagulation disorders other than haemophilia B
* Previous arterial thrombotic events (e.g. myocardial infarction and intracranial thrombosis) or previous deep venous thrombosis or pulmonary embolism (as defined by available medical records)
* Any disease (liver, kidney, inflammatory and mental disorders included) or condition which, according to the Investigator's (trial physician) judgement, could imply a potential hazard to the patient, interfere with trial participation, or interfere with trial outcome

Ages: 13 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2012-04-15 (Actual); Primary Completion 2014-03-30 (Actual); Study Completion 2014-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (48):
- United States (13):
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, San Francisco, California
  - Novo Nordisk Investigational Site, Washington D.C., District of Columbia
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Augusta, Georgia
  - Novo Nordisk Investigational Site, Iowa City, Iowa
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Omaha, Nebraska
  - Novo Nordisk Investigational Site, Newark, New Jersey
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, Houston, Texas
- Novo Nordisk Investigational Site, Vienna, Austria
- France (2):
  - Novo Nordisk Investigational Site, Bron
  - Novo Nordisk Investigational Site, Le Kremlin-Bicêtre
- Germany (4):
  - Novo Nordisk Investigational Site, Bonn
  - Novo Nordisk Investigational Site, Duisburg
  - Novo Nordisk Investigational Site, Giessen
  - Novo Nordisk Investigational Site, Hanover
- Novo Nordisk Investigational Site, Athens, Greece
- Italy (2):
  - Novo Nordisk Investigational Site, Florence
  - Novo Nordisk Investigational Site, Milan
- Japan (6):
  - Novo Nordisk Investigational Site, Kashihara-shi, Nara
  - Novo Nordisk Investigational Site, Kawasaki-shi, Kanagawa
  - Novo Nordisk Investigational Site, Nagoya-shi, Aichi
  - Novo Nordisk Investigational Site, Nishinomiya-shi
  - Novo Nordisk Investigational Site, Shinjuku-ku, Tokyo
  - Novo Nordisk Investigational Site, Suginami-ku, Tokyo
- Novo Nordisk Investigational Site, Kuala Lumpur, Malaysia
- Novo Nordisk Investigational Site, Utrecht, Netherlands
- Novo Nordisk Investigational Site, Skopje, North Macedonia
- Novo Nordisk Investigational Site, Timișoara, Timiș County, Romania
- Russia (2):
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Saint Petersburg
- Novo Nordisk Investigational Site, Parktown Johannesburg, Gauteng, South Africa
- Spain (2):
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Valencia
- Novo Nordisk Investigational Site, Taipei, Taiwan
- Novo Nordisk Investigational Site, Bangkok, Thailand
- Turkey (Türkiye) (3):
  - Novo Nordisk Investigational Site, Ankara
  - Novo Nordisk Investigational Site, Kayseri
  - Novo Nordisk Investigational Site, Konya
- United Kingdom (5):
  - Novo Nordisk Investigational Site, Basingstoke
  - Novo Nordisk Investigational Site, Cardiff
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, Manchester
  - Novo Nordisk Investigational Site, Oxford

REFERENCES:
- [Background] Young G, Collins P, Tehranchi R, Chuansumrit A, Hanabusa H, Lentz SR, Mahlangu J, Mauser-Bunschoten E, Negrier C, Oldenburg J, Patiroglu T, Santagostino E, Zak M, Abdul Karim F. Safety and efficacy of nonacog beta pegol (N9-GP) for prophylaxis and treatment of bleeding episodes in previously-treated patients with hemophilia B: results from an extension trial. American Society of Hematology - 56th Annual Meeting (ASH) in San Francisco, CA, US
- [Result] Young G, Collins PW, Colberg T, Chuansumrit A, Hanabusa H, Lentz SR, Mahlangu J, Mauser-Bunschoten EP, Negrier C, Oldenburg J, Patiroglu T, Santagostino E, Tehranchi R, Zak M, Karim FA. Nonacog beta pegol (N9-GP) in haemophilia B: A multinational phase III safety and efficacy extension trial (paradigm4). Thromb Res. 2016 May;141:69-76. doi: 10.1016/j.thromres.2016.02.030. Epub 2016 Mar 2. PMID 26970716
- [Result] Chowdary P, Kearney S, Regnault A, Hoxer CS, Yee DL. Improvement in health-related quality of life in patients with haemophilia B treated with nonacog beta pegol, a new extended half-life recombinant FIX product. Haemophilia. 2016 Jul;22(4):e267-74. doi: 10.1111/hae.12995. Epub 2016 Jun 28. PMID 27352908
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 41 sites in 15 countries as follows: France: 1 site; Germany: 3 sites; Italy: 2 sites; Japan: 4 sites; Macedonia: 2 sites; Malaysia: 1 site; Netherlands: 1 site; Romania: 1 site, Russia: 1 site; South Africa: 1 site; Taiwan: 1 site, Thailand: 2 sites; Turkey: 3 sites; United Kingdom: 5 sites; United States: 13 sites
Pre-assignment Details: A total of 71 unique subjects were dosed during this trial. During the trial, subjects were free to switch between treatment arms if agreed between the investigator and the subject. Subjects who switched arms were represented in multiple arms.
Groups:
- Prophylaxis 10 IU/kg: Subjects were given 10 IU/kg weekly nonacog beta pegol. Subjects were free to switch between treatment arms if agreed between the investigator and the subject. Administration of the appropriate volume of nonacog beta pegol was given as an intravenous (i.v.) bolus injection. The maximum injection rate was 4 mL/min. Subjects on prophylaxis who experienced a bleeding episode were to treat the bleeding episode with a single dose of 40 IU/kg, unless the bleeding episode was severe in which case it was to be treated with 80 IU/kg.
- Prophylaxis 40 IU/kg: Subjects were given 40 IU/kg weekly nonacog beta pegol. Subjects were free to switch between treatment arms if agreed between the investigator and the subject. Administration of the appropriate volume of nonacog beta pegol was given as an i.v. bolus injection. The maximum injection rate was 4 mL/min. Subjects on prophylaxis who experienced a bleeding episode were to treat the bleeding episode with a single dose of 40 IU/kg, unless the bleeding episode was severe in which case it was to be treated with 80 IU/kg.
- Prophylaxis 80 IU/kg: Subjects were dosed with 80 IU/kg every second week. Subjects were free to switch between treatment arms if agreed between the investigator and the subject. Administration of the appropriate volume of nonacog beta pegol was given as an i.v. bolus injection. The maximum injection rate was 4 mL/min. Subjects on prophylaxis who experienced a bleeding episode were to treat the bleeding episode with a single dose of 40 IU/kg, unless the bleeding episode was severe in which case it was to be treated with 80 IU/kg.
- On-demand: Subjects in the on-demand group were administered with the single dose of 40 IU/kg of nonacog beta pegol. The recommended dose for treatment of a mild or moderate bleeding episode, for example a joint bleed, was a single dose of 40 IU/kg nonacog beta pegol. If there was no observed effect of 40 IU/kg, the investigator was to be contacted prior to administration of the second dose of 40 IU/kg. The recommended dose for severe bleeds was 80 IU/kg nonacog beta pegol. Subjects were free to switch between treatment arms if agreed between the investigator and the subject.
Period: Overall Study
Arm/Group | Prophylaxis 10 IU/kg | Prophylaxis 40 IU/kg | Prophylaxis 80 IU/kg | On-demand
Started | 18 | 48 | 0 | 5
After Switching the Arms (Patients were free to switch between treatment arms if agreed between investigator and patient) | 21 (18 subjects started in this arm and additional 3 subjects from 40 IU/kg switched to this arm) | 52 (48 subjects started in this arm, 3 subjects in 10 IU/kg+1 subject in on-demand switched to this arm) | 2 (No subjects started in this arm initially, 2 patients in 40 IU/kg arm switched to this arm.) | 5
Completed | 16 | 44 | 0 | 5
Not Completed | 2 | 4 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Withdrawal criteria | 0 | 2 | 0 | 0
Not completed — Unclassified | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) consisted of all subjects exposed to nonacog beta pegol.
Groups:
- Prophylaxis 10 IU/kg: Subjects were given 10 IU/kg weekly nonacog beta pegol. Subjects were free to switch between treatment arms if agreed between the investigator and the subject. Administration of the appropriate volume of nonacog beta pegol was given as an i.v. bolus injection. The maximum injection rate was 4 mL/min. Subjects on prophylaxis who experienced a bleeding episode were to treat the bleeding episode with a single dose of 40 IU/kg, unless the bleeding episode was severe in which case it was to be treated with 80 IU/kg.
- Total: Total of all reporting groups
Arm/Group | Prophylaxis 10 IU/kg | Prophylaxis 40 IU/kg | Prophylaxis 80 IU/kg | On-demand | Total
Number analyzed (Participants) | 18 | 48 | 0 | 5 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.2 (13.6) | 31.4 (14.4) |  | 37.6 (15.4) | 32.0 (14.2)
Age, Customized [Number; unit: Participants]
  13 - 17 years | 3 | 12 |  | 0 | 15
  18 - 70 years | 15 | 36 |  | 5 | 56
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 18 | 48 | 0 | 5 | 71

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Inhibitory Antibodies Against FIX Defined as Titre Above or Equal to 0.6 BU (Bethesda Units)
Description: The primary endpoint was incidence of inhibitors against coagulation factor nine (FIX) defined as titre
  ≥0.6 Bethesda unit (BU). Number of subjects who developed inhibitors against FIX are reported.
Time Frame: From Day 1 up to 2 years
Population: Safety Analysis Set consisted of all subjects exposed to nonacog beta pegol. Subjects who switched arms were represented in multiple columns.
Measure: Number; unit: Patients with inhibitory antibodies
Arm/Group | Prophylaxis 10 IU/kg | Prophylaxis 40 IU/kg | Prophylaxis 80 IU/kg | On-demand
Number analyzed (Participants) | 21 | 52 | 2 | 5
Patients with inhibitory antibodies | 0 | 0 | 0 | 0

2. Secondary Outcome: Haemostatic Effect of Nonacog Beta Pegol When Used for Treatment of Bleeding Episodes, Assessed as Success/Failure Based on a Four-point Scale for Haemostatic Response (Excellent, Good, Moderate, Poor)
Description: The haemostatic effect was evaluated by a four-point scale where an "excellent" or "good" outcome translated into a successful treatment, and a "moderate" or "poor" outcome was considered a treatment failure. The values mentioned below do not include bleeds with missing response.
Time Frame: From Day 1 up to 2 years
Population: Full analysis set consisted of all subjects exposed to nonacog beta pegol. Subjects who switched arms were represented in multiple columns.
Measure: Number; unit: Percentage of bleeding episodes
Units Other Than Participants: Bleeding episodes
Groups:
- Total: Subjects received nonacog beta pegol as prophylaxis treatment or on-demand treatment. Subjects in the prophylaxis treatment received either 10 IU/kg once weekly, 40 IU/kg once weekly or 80 IU/kg once every second week. Subjects in the on-demand group were administered with a single dose of 40 IU/kg of nonacog beta pegol. Subjects with on-demand treatment and prophylaxis treatments who experienced a bleeding episode were to be treated with single dose of 40 IU/kg unless the bleeding episode was severe in which case it was to be treated with 80 IU/kg. Administration of the appropriate volume of nonacog beta pegol was given as an i.v. bolus injection. The maximum injection rate was 4 mL/min. Subjects were free to switch between treatment arms if agreed between the investigator and the subject.
Arm/Group | Prophylaxis 10 IU/kg | Prophylaxis 40 IU/kg | Prophylaxis 80 IU/kg | On-demand | Total
Number analyzed (Participants) | 21 | 52 | 2 | 5 | 71
Number analyzed (Bleeding episodes) | 35 | 98 | 1 | 73 | 207
Percentage of bleeding episodes
  Success | 97.1 | 94.8 | 100 | 93.2 | 94.6
  Failure | 2.9 | 5.2 | 0 | 6.8 | 5.4

3. Secondary Outcome: Number of Bleeding Episodes During Routine Prophylaxis
Description: Annualized bleeding rate is the total number of bleeding episodes/total exposure time. It is analysed by a Poisson regression model with dose as a factor allowing for over-dispersion and using treatment duration as an offset. Median annualized bleeding rate is the median of individual annualized bleeding rates. Numbers are based on the treatment arm at the time of each bleed.
Time Frame: From Day 1 up to 2 years
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: bleeds/patient/year
Arm/Group | Prophylaxis 10 IU/kg | Prophylaxis 40 IU/kg | Prophylaxis 80 IU/kg
Number analyzed (Participants) | 21 | 52 | 2
bleeds/patient/year | 1.36 [0.00 to 2.23] | 1.00 [0.00 to 2.03] | 0 [0 to 0]

4. Secondary Outcome: FIX Trough Levels
Description: During the trial, the pre-dose FIX levels was measured with the one-stage clotting assay. Measurements taken at least 5 days and no more than 10 days after last dose as well as at least 14 days after last bleeding episode were included in this analysis. The mean FIX trough levels were estimated based on the mixed effects model on the log-transformed plasma concentration with subject as a random effect. The mean FIX trough level was presented back-transformed to the natural scale.
Time Frame: From Day 1 up to 2 years
Population: Full analysis set consisted of all subjects exposed to nonacog beta pegol. This endpoint was analysed only for the prophylaxis arms (i.e.,10 IU/kg, 40 IU/kg). No pre-dose measurements were collected for patients on 80 IU/kg every second week prophylaxis.
Measure: Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Prophylaxis 10 IU/kg | Prophylaxis 40 IU/kg
Number analyzed (Participants) | 21 | 52
IU/mL | 0.098 [0.080 to 0.119] | 0.213 [0.189 to 0.241]

5. Secondary Outcome: Incidence of Adverse Events (AEs)
Description: AEs were summarized by frequency of events and frequency of patients with any event. Incidence of AEs was expressed as number of AEs per subject years of exposure (total number of events /total time in trial).
Time Frame: From Day 1 up to 2 years
Population: Safety Analysis Set consisted of all subjects who were exposed to nonacog beta pegol. Subjects who switched arms were represented in multiple columns.
Measure: Number; unit: Events per subject year of exposure
Arm/Group | Prophylaxis 10 IU/kg | Prophylaxis 40 IU/kg | Prophylaxis 80 IU/kg | On-demand
Number analyzed (Participants) | 21 | 52 | 2 | 5
Events per subject year of exposure | 2.4 | 1.9 | 0 | 3.2

6. Secondary Outcome: Incidence of Serious Adverse Events (SAEs)
Description: AEs were summarized by frequency of events and frequency of patients with any event. Incidence of serious AEs was expressed as number of serious AEs per subject years of exposure (total number of events /total time in trial).
Time Frame: From Day 1 up to 2 years
Population: as for outcome 1
Measure: Number; unit: Events per subject year of exposure
Arm/Group | Prophylaxis 10 IU/kg | Prophylaxis 40 IU/kg | Prophylaxis 80 IU/kg | On-demand
Number analyzed (Participants) | 21 | 52 | 2 | 5
Events per subject year of exposure | 0.1 | 0.1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) from baseline visit (visit 1) and until one week after last treatment with nonacog beta pegol (±2 days) (up to 2 years)
Description: The safety analysis set consists of all patients exposed to nonacog beta pegol.
Groups:
- Prophylaxis 10 U/kg: Subjects were given 10 IU/kg weekly nonacog beta pegol. Subjects were free to switch between treatment arms if agreed between the investigator and the subject. Administration of the appropriate volume of nonacog beta pegol was given as an intravenous (i.v.) bolus injection. The maximum injection rate was 4 mL/min. Subjects on prophylaxis who experienced a bleeding episode were to treat the bleeding episode with a single dose of 40 IU/kg, unless the bleeding episode was severe in which case it was to be treated with 80 IU/kg.
- Prophylaxis 40 U/kg: Subjects were given 40 IU/kg weekly nonacog beta pegol. Subjects were free to switch between treatment arms if agreed between the investigator and the subject. Administration of the appropriate volume of nonacog beta pegol was given as an i.v. bolus injection. The maximum injection rate was 4 mL/min. Subjects on prophylaxis who experienced a bleeding episode were to treat the bleeding episode with a single dose of 40 IU/kg, unless the bleeding episode was severe in which case it was to be treated with 80 IU/kg.
- Prophylaxis 80 U/kg: Subjects were dosed with 80 IU/kg every second week. Subjects were free to switch between treatment arms if agreed between the investigator and the subject. Administration of the appropriate volume of nonacog beta pegol was given as an i.v. bolus injection. The maximum injection rate was 4 mL/min. Subjects on prophylaxis who experienced a bleeding episode were to treat the bleeding episode with a single dose of 40 IU/kg, unless the bleeding episode was severe in which case it was to be treated with 80 IU/kg.
Arm/Group | Prophylaxis 10 U/kg | Prophylaxis 40 U/kg | Prophylaxis 80 U/kg | On-demand
Serious Adverse Events (participants affected / at risk) | 1/21 | 5/52 | 0/2 | 0/5
Other Adverse Events (participants affected / at risk) | 8/21 | 8/52 | 0/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylaxis 10 U/kg (N=21) | Prophylaxis 40 U/kg (N=52) | Prophylaxis 80 U/kg (N=2) | On-demand (N=5)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prophylaxis 10 U/kg (N=21) | Prophylaxis 40 U/kg (N=52) | Prophylaxis 80 U/kg (N=2) | On-demand (N=5)
Asthenopia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 4 (6) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 3 (5) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (5) | 4 (5) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.